CLINICAL TRIAL: NCT05169892
Title: Canadian Cohort of Aquablation, a Robotically Executed, Surgeon-guided, High-pressure Water Jet Ablation Therapy for Endoscopic Resection of Prostate Tissue, in Benign Prostatic Hyperplasia (BPH).
Brief Title: Aquablation in Benign Prostatic Hyperplasia in Canada
Status: Recruiting | Type: Observational
Sponsor: Can-Am HIFU Inc. (Other)
Responsible Party: Principal Investigator, Dean Elterman, Urologist, Can-Am HIFU Inc.
Other Study IDs: Aquablation in BPH
Record Dates: First submitted 2021-11-27; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Urologic Diseases
Keywords: benigh prostate hypertrophy
MeSH Terms: conditions — Urologic Diseases | interventions — Aquablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aquablation
  Interventions: Procedure: Aquablation

INTERVENTIONS:
Procedure: Aquablation — Aquablation

SUMMARY:
To document the clinical outcome of Aquablation therapy for BPH patient in Canadian cohort.

DETAILED DESCRIPTION:
Patients will be followed up for 3 years as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Benign Prostate Hypertrophy (BPH)
* Male subjects of ≥ 18 years of age
* Candidate for Aquablation therapy as per clinical decision of Investigator
* Willing and able to accurately complete questionnaires
* Willing and able to provide signed and dated informed consent

Exclusion Criteria:

* Characteristics indicating a poor compliance with study protocol requirements.
* Disease or other health condition that is not suitable for this study.
* Unable or unwilling to provide signed informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BPH patients treated by Aquablation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum flow rate (Q-max) | Baseline
  Standard of care
Post-Void Residual (PVR) volume | Baseline
  Standard of care
Maximum flow rate (Q-max) | 1 month after surgery
  Standard of care
Post-Void Residual (PVR) volume | 1 month after surgery
  Standard of care
Maximum flow rate (Q-max) | 3 months after surgery
  Standard of care
Post-Void Residual (PVR) volume | 3 months after surgery
  Standard of care
Maximum flow rate (Q-max) | 6 months after surgery
  Standard of care
Post-Void Residual (PVR) volume | 6 months after surgery
  Standard of care
Maximum flow rate (Q-max) | 12 months after surgery
  Standard of care
Post-Void Residual (PVR) volume | 12 months after surgery
  Standard of care
Maximum flow rate (Q-max) | 24 months after surgery
  Standard of care
Post-Void Residual (PVR) volume | 24 months after surgery
  Standard of care
Maximum flow rate (Q-max) | 36 months after surgery
  Standard of care
Post-Void Residual (PVR) volume | 36 months after surgery
  Standard of care
Prostate Volume | Baseline
  Standard of care
Prostate Volume | 12 months after surgery
  Standard of care
Questionnaires | Baseline
  IPSS
Questionnaires | 1 month after surgery
  IPSS
Questionnaires | 3 months after surgery
  IPSS
Questionnaires | 6 months after surgery
  IPSS
Questionnaires | 12 months after surgery
  IPSS
Questionnaires | 24 months after surgery
  IPSS
Questionnaires | 36 months after surgery
  IPSS
Adverse Events | Baseline
  Adverse Events
Adverse Events | 1 day of Surgery
  Adverse Events
Adverse Events | 1 month after surgery
  Adverse Events
Adverse Events | 3 months after surgery
  Adverse Events
Adverse Events | 6 months after surgery
  Adverse Events
Adverse Events | 12 months after surgery
  Adverse Events
Adverse Events | 24 months after surgery
  Adverse Events
Adverse Events | 36 months after surgery
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Dean Elterman, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No